CLINICAL TRIAL: NCT04665830
Title: PCSK 9 Inhibition as Secondary Prevention in Renal Transplant Patients With Cardiovascular Disease.
Brief Title: PCSK 9 Inhibition as Secondary Prevention in Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamid Al-Essa Organ Transplant Center (Other Government)
Responsible Party: Principal Investigator, Osama Gheith, Consultant nephrologist, Hamid Al-Essa Organ Transplant Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/789
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Kideny Transplant Recipients With High Cardiovascular Risk Score
MeSH Terms: interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: all renal transplant recipients who are followed up in Hamed Al-Essa organ transplant center of Kuwait for 6 months duration. Cardio-vascular risk score will be estimated using the Framingham score. Patients with scores higher than 10 will be randomized in this prospective controlled study to receive either the evolocumab (group 1, n=100 patients) or the conventional group (group 2, n=100 patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Evolocumab group, patients who are receiving this therapy for 12 months.
  Interventions: Drug: Evolocumab
- Group 2 (Placebo Comparator): The Statin group includes patients who are maintained on statin therapy.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — treated patients with evolocumab for high cholesterol

SUMMARY:
From this randomized controlled study, we aim to:

A.Do do cardiovascular risk stratification of renal transplant recipients who are followed up in Hamed Al-Essa organ transplant center of Kuwait.

B. To compare the effectiveness of a PCSK9 inhibitor plus maximum tolerated statin therapy vs. maximum tolerated statin therapy alone in the reduction of major cardiovascular events among renal transplant recipients with cardiovascular disease.

C. To compare the effectiveness of a PCSK9 inhibitor plus maximum tolerated statin therapy vs. maximum tolerated statin therapy alone in terms of LDL-C-lowering, muscle symptoms, and quality of life.

D. To compare patient adherence to the different treatment protocols.

DETAILED DESCRIPTION:
Background:

Low-density lipoprotein (LDL) cholesterol is a well-established and modifiable risk factor for cardiovascular disease. Monoclonal antibodies that inhibit proprotein convertase subtilisin-kexin type 9 (PCSK9) have emerged as a new class of drugs that effectively lower LDL cholesterol levels.1 Approximately 735,000 Americans have a myocardial infarction each year (2), and about 800,000 have a stroke. (3) Many patients remain at increased cardiovascular risk despite maximum tolerated statin therapy and could benefit from further LDL-C reduction. Most patients are treated with HMG-CoA reductase inhibitors, commonly known as statins. Millions of patients are eligible for cholesterol-lowering medication, according to current guidelines.4 High-intensity statin therapy reduces LDL-C and cardiovascular events more than moderate intensity statin therapy. 5 However, the response to statins is variable, and in some patients it is not tolerable (between 7 percent and 29 percent of patients taking statins report having muscle symptoms) 6, which represent a principal reason for nonadherence. Moreover, high-intensity statin therapy may have less benefit in low-risk primary prevention patients with a modest increase in the incidence of diabetes in such cases 5, 7. Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors are currently indicated for some patients at high risk, including those with familial hypercholesterolemia or pre-existing cardiovascular disease. PCSK9 inhibitors are a new class of medications that have been found to be very effective in reducing LDL-C, either as monotherapy or when added to background statin therapy. Normally, PCSK9 binds to low-density lipoprotein cholesterol (LDL-C) receptors, reducing the activity of the LDL-C receptors. PCSK9 inhibitors prevent PCSK9 from binding to the LDL receptor, thereby increasing the activity of the receptors and enhancing removal of LDL-C from circulation. 8 Current guidelines recommend that patients whose 10-year risk of major cardiovascular events is 10 percent or greater take statins. 9 Two PCSK9 inhibitors are currently available and approved by FDA for use in the United States: evolocumab and alirocumab. These drugs are monoclonal antibodies (mAbs) administered by Proposed Clinical Trial Protocol on Use of PCSK9 Inhibitors for Primary Prevention of Cardiovascular Disease 3 subcutaneous injection bi-weekly or monthly and are currently approved for patients with familial hypercholesterolemia or clinical atherosclerotic cardiovascular disease who require additional lowering of LDL-C. Two recent reports on the effects of evolocumab and alirocumab have raised expectations that these drugs will dramatically reduce cardiovascular events.10,11 the rate of major cardiovascular events was lower with alirocumab than with placebo (1.7 percent versus 3.3 percent; hazard ratio 0.52; 95 percent confidence interval 0.31 to 0.90; P=0.02). 11 Notably, the annual cost for a single patient in the United States for PCSK9 inhibitors is approximately $14,000.9 The prevalence of cardiovascular diseases (CVD) has increased in kidney transplant recipients. CVD remains a leading cause of mortality among recipients with functioning grafts. The pathophysiology of CVD recipients is a complex interplay between preexisting risk factors, metabolic sequelae of immunosuppressive agents, infection, and rejection.17

Aim of the study:

A. Cardiovascular risk stratification of renal transplant recipients who are followed up in Hamed Al-Essa organ transplant center of Kuwait.

B. To compare the effectiveness of a PCSK9 inhibitor plus maximum tolerated statin therapy vs. maximum tolerated statin therapy alone in the reduction of major cardiovascular events among renal transplant recipients with cardiovascular disease.

C. To compare the effectiveness of a PCSK9 inhibitor plus maximum tolerated statin therapy vs. maximum tolerated statin therapy alone in terms of LDL-C-lowering, muscle symptoms, and quality of life.

D. To compare patient adherence to the different treatments protocols.

Patient and methods:

Patients eligible for participation in this study are renal transplant recipients aged between 30 and 80 years and have clinically evident atherosclerotic cardiovascular disease, defined as a history of myocardial infarction, non-hemorrhagic stroke, or symptomatic peripheral artery disease, as well as additional characteristics that placed them at higher cardiovascular risk.

This group of patients will be selected after screening of all renal transplant recipients who are followed up in Hamed Al-Essa organ transplant center of Kuwait along 6 months duration. Cardio-vascular risk score will be estimated using Framingham score. Patients with score higher than 20 will be randomized in this prospective controlled study to receive either the evolocumab (group 1, n=100 patients) or the conventional group (group 2, n=100 patients).

The selection criteria:

1. Signed informed consent, 2. Male or female Kuwaiti older than 30 and younger than ≤ 80 years of age at signing of informed consent 3. History of clinically evident cardiovascular disease(diagnosis of myocardial infarction ; non-hemorrhagic stroke or symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with ankle-brachial index (ABI) < 0.85, or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease, 4. At least 1 major risk factor or at least 2 minor risk factors below: Major Risk Factors (1 Required): o diabetes (type 1 or type 2) o age ≥ 65 years at randomization (and ≤ 85 years at time of informed consent) o MI or non-hemorrhagic stroke within 6 months of screening o additional diagnosis of myocardial infarction or non-hemorrhagic stroke excluding qualifying MI or non-hemorrhagic stroke o current daily cigarette smoking o history of symptomatic PAD (as mentioned before) if eligible by MI or stroke history; Minor Risk Factors (2 Required): o history of non-MI related coronary revascularization o residual coronary artery disease with ≥ 40% stenosis in ≥ 2 large vessels o Most recent HDL-C <1.0 mmol/L for men and <1.3 mmol/L for women by central laboratory before randomization o Most recent CRP > 2.0 mg/L by central laboratory before randomization o Most recent LDL-C ≥ 3.4 mmol/L or non-HDL-C ≥ 4.1 mmol/L by central laboratory before randomization o metabolic syndrome.

Exclusion Criteria:

1. Recent MI or stroke 2. NYHA class III or IV, or last known left ventricular ejection fraction < 30% 3. Known hemorrhagic stroke at any time 4. Uncontrolled or recurrent ventricular tachycardia 5. Planned or expected cardiac surgery or revascularization within 3 months after randomization 6. Uncontrolled hypertension (sitting systolic blood pressure (SBP) > 180 mmHg or diastolic BP (DBP) > 110 mmHg), 7. Prior use of PCSK9 inhibition treatment other than evolocumab or use of evolocumab < 12 weeks prior to final lipid screening 8. Untreated or inadequately treated hyperthyroidism or hypothyroidism (thyroid stimulating hormone (TSH) < lower limit of normal or > 1.5 times the upper limit of normal and free thyroxine (T4) levels that are outside normal range at final screening. ,9. Severe renal graft dysfunction(estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2 at final screening, 10. Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN as determined by central laboratory analysis at final screening. 11. Personal or family history of hereditary muscular disorders. 12. Malignancy or HIV patients, 13. Known major active infection or major hematologic, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator, 13. Female subject who has either (1) not used acceptable method(s) of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment with IP and for an additional 15 weeks after the end of treatment with IP, unless the subject is sterilized or postmenopausal; 23. Known sensitivity to any of the active substances or their excipients to be administered during dosing.

Methods:

The baseline characteristics of the patients in the two groups will be collected with special stress on demographic data, history of myocardial infarction, history of previous non-hemorrhagic stroke, and symptomatic peripheral artery disease. At baseline, all patients will be on statin therapy (defined in accordance with American College of Cardiology and American Heart Association joint guidelines12) and or ezetimibe. All antihypertensive medications, antiplatelet and diuretic therapy will be recorded. The duration of follow-up will be 12 months.

Randomization:

Eligible patients will be randomly assigned in a 1:1 ratio to receive subcutaneous injections of evolocumab (either 140 mg every 2 weeks) or matching placebo. Randomization will be performed in a double-blinded manner with the use of a central computerized system, with stratification according to the final screening LDL cholesterol level (<2.2 or ≥2.2 mmol per liter) and region.

Follow up:

All patients will be followed up in Hamed Al-Essa organ transplant center clinics at least every 2 months or according the local follow up protocol. Patients who have a fasting LDL cholesterol level of 1.8 mmol per liter or higher or a non-high-density lipoprotein (HDL) cholesterol level of 2.6 mmol per liter or higher while they were taking an optimized regimen of lipid-lowering therapy, which was defined as preferably a high intensity statin but must have been at least atorvastatin at a dose of 20 mg daily with or without ezetimibe.

Our immunosuppression protocol consists of 5 doses of antithymocyte globulin (Sanofi US, Bridgewater, NJ, USA) for high risk patients (as re-transplants, prior pregnancy, blood transfusion, HLA-antibody positive and or more than 4 HLA mismatches)or 2 doses of IL-2 receptor blocker (basiliximab; Novartis, Inc., Switzerland) for low risk patients. Maintenance therapy consists of prednisolone, MMF and a calcineurin inhibitor (CNI). The dose of CNI will be gradually decreasing till the lowest dose by the end of the 1st year guided by 12-hour trough level. We keep the cyclosporine A level between 200 to 250 ng/ml during 1st month then between 150-200 ng/ml for a couple of months then between 125-150 ng/ml for 2 months and from 75-125 ng/ml till the end of the 1st year. Similarly, we keep tacrolimus trough levels between 8 to 10 ng/ml during 1st 3 months then from 5-8 ng/ml thereafter. Maintenance immunosuppression with sirolimus based regimen will be used to rejection free patients with low immunological risk after 3 months of transplantation.

Acute cellular rejection (ACR) will be treated with intravenous methylprednisolone sodium succinate (solumedrol 1 gram daily for 3 days) and or thymoglobulin (1 mg /kg for 7 -10 days) for steroid resistant rejection. Antibody mediated rejection (AAMR) will be treated with plasma exchange, IVIG (2gm/kg) and rituximab. Patients, who will receive thymoglobulin as antirejection, will be managed by secondary prophylaxis for 1 month. Patients will be monitored daily during hospital stay then at each outpatient visit with complete blood picture, serum creatinine, creatinine clearance, liver function tests (bilirubin, liver enzymes and albumin) and drug levels.

Lipid Data:

The LDL cholesterol level will be checked in the central laboratory for all patients in both groups at baseline (according to routine laboratory analysis) and every third month using desktop Mission CE0123 cholesterol monitoring machine, till the end of the study.

End Points:

The primary efficacy end point will be any major cardiovascular events, defined as the cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization. The key secondary efficacy end point will be cardiovascular death, myocardial infarction, or stroke. Safety was assessed through collection of data on adverse events and central laboratory testing in Ibn Sina laboratory, Sabah area of Kuwait.

Statistics and sample size calculation:

Statistical analysis of data will be evaluated on computer using SPSS (Statistical Package for Social Science for Windows) 11.0 package software (SPSS Inc., Chicago, IL, USA). In order to analyze the identifying and disease related characteristics of patients, matched t-test will be used to compare means and standard deviations of numerical variables of the two groups and to test whether there will be a difference between pre-education and post-education score averages. Categorical data will be compared using the chi square test. Values for P less than .05 were considered significant.

Confidentiality and consent :

To maintain confidentiality, all research data, blood and/urine specimens, Consent Forms, Data Collection Forms, reports, and other records that leave the site will be identified only by a Code Number-participant identification number (Participant ID). All records will be kept in a locked file cabinet. All computer entry and networking programs will be done using PIDs only. Participants' identifiable private information will not be released to a third party without written permission of the participants.

Detailed information will be delivered to each patient about the study including the aim and benefits. Before starting the enrolment of each patient, the investigator will get signed informed consent which will be kept in patient file. Moreover, a copy of this consent will be given to the patient.

* We will exclude participants with diminished capacity, such as minors and mentally retarded, who cannot consent for themselves from this study.
* The original copy of the consent will be kept in the investigators' records, a copy will be given to each participant, and this will be documented in the participant's record.
* The primary investigator and co-primary investigators will be responsible for implementing the consenting process and obtaining the Informed Consent of Participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent, 2. Male or female Kuwaiti older than 30 and younger than ≤ 80 years of age at the signing of informed consent 3. History of clinically evident cardiovascular disease(diagnosis of myocardial infarction; non-hemorrhagic stroke or symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with the ankle-brachial index (ABI) < 0.85, or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease, 4. At least 1 major risk factor or at least 2 minor risk factors below: Major Risk Factors (1 Required): o diabetes (type 1 or type 2) o age ≥ 65 years at randomization (and ≤ 85 years at the time of informed consent) o MI or non-hemorrhagic stroke within 6 months of screening o additional diagnosis of myocardial infarction or non-hemorrhagic stroke excluding qualifying MI or non-hemorrhagic stroke o current daily cigarette smoking o history of symptomatic PAD (as mentioned before) if eligible by MI or stroke history; Minor Risk Factors (2 Required): o history of non-MI related coronary revascularization o residual coronary artery disease with ≥ 40% stenosis in ≥ 2 large vessels o Most recent HDL-C <1.0 mmol/L for men and <1.3 mmol/L for women by the central laboratory before randomization o Most recent CRP > 2.0 mg/L by the central laboratory before randomization o Most recent LDL-C ≥ 3.4 mmol/L or non-HDL-C ≥ 4.1 mmol/L by the central laboratory before randomization o metabolic syndrome.

Exclusion Criteria:

* Exclusion Criteria:

  1. Recent MI or stroke 2. NYHA class III or IV, or last known left ventricular ejection fraction < 30% 3. Known hemorrhagic stroke at any time 4. Uncontrolled or recurrent ventricular tachycardia 5. Planned or expected cardiac surgery or revascularization within 3 months after randomization 6. Uncontrolled hypertension (sitting systolic blood pressure (SBP) > 180 mmHg or diastolic BP (DBP) > 110 mmHg), 7. Prior use of PCSK9 inhibition treatment other than evolocumab or use of evolocumab < 12 weeks prior to final lipid screening 8. Untreated or inadequately treated hyperthyroidism or hypothyroidism (thyroid-stimulating hormone (TSH) < lower limit of normal or > 1.5 times the upper limit of normal and free thyroxine (T4) levels that are outside normal range at the final screening. ,9. Severe renal graft dysfunction(estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2 at final screening, 10. Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN as determined by central laboratory analysis at the final screening. 11. Personal or family history of hereditary muscular disorders. 12. Malignancy or HIV patients, 13. Known major active infection or major hematologic, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator, 13. Female subject who has either (1) not used-acceptable method(s) of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment with IP and for an additional 15 weeks after the end of treatment with IP unless the subject is sterilized or postmenopausal; 23. Known sensitivity to any of the active substances or their excipients to be administered during dosing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Any major cardiovascular events | 24 months
  cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- OTC, MOH , Kuwait, Kuwait City, Kuwait